CLINICAL TRIAL: NCT00302484
Title: Use of Bisphosphonates in the Treatment of Osteopathy After Liver Transplantation, a Prospective Randomised Study
Brief Title: Use of Bisphosphonates in the Treatment of Osteopathy After Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LTX-BISPHO-01
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2006-07-26 (Estimated); Status verified 2006-01

CONDITIONS: Osteoporosis; Liver Transplantation
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronate

SUMMARY:
Patients with a terminal chronic liver disease have a disordered bone metabolism resulting in a higher risk of falling ill with osteoporosis. Although liver transplantation restores liver function, immunosuppressive therapy (especially corticosteroids) after transplantation increases again the risk of osteoporosis and bone fragility. Zoledronate, a bisphosphonate, slows down the destruction of bone. The purpose of this study is to determine whether bisphosphonates are effective in the prevention of osteoporosis following immunosuppressive therapy after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* primary liver transplantation
* retransplantation within two weeks
* written informed consent
* Age ≥ 18 years

Exclusion Criteria:

* chronic kidney disease:
* Creatinine Clearance < 35 ml/min or Serum Creatinine > 2,5 mg/dl
* known hypersensitivity to Zoledronate, or any of the recipients of the drug
* bone specific medication (Bisphosphonate, Fluoride, Calcitonin) within the last three months before liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96
Dates: Start 2002-04

PRIMARY OUTCOMES:
first bone fracture or death within 24 months after liver transplantation

SECONDARY OUTCOMES:
bone mineral density (pre-transplant, 6 and 12 months post-transplant)
serum biochemical bone markers (osteocalcin, alkaline phosphatase, parathyroid hormone)
histomorphometric measurements of transiliacal bone biopsies (intraoperative, 6 months post-transplant)

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Mühlbacher, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Surgery, Division of Transplantation, Vienna, Vienna, Austria